CLINICAL TRIAL: NCT02744664
Title: A Single Arm, Open Label, Perspective Study to Determine the Efficacy and Safety of Icotinib Combine Cryotherapy for Advanced NSCLC Patients
Brief Title: Cryotherapy Combine Icotinib for Advanced NSCLC Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUDA2016004
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Lung Neoplasms
Keywords: Lung Neoplasms; EGFR mutation; Cryotherapy; Icotinib
MeSH Terms: conditions — Lung Neoplasms | interventions — Cryotherapy; Cryosurgery; icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): The subject receive Cryotherapy and than receive Icotinib 125mg, 3 times a day, orally administered until disease progression or intolerable toxicity reaction.
  Interventions: Procedure: Cryotherapy; Drug: Icotinib

INTERVENTIONS:
Procedure: Cryotherapy — After entering the group subject receive Cryotherapy on lung cancer
  Other Names: Cryoablation
Drug: Icotinib — After Cryotherapy, subjects begin Icotinib administration
  Other Names: EGFR-TKI

SUMMARY:
This trial is to designed to assess the efficacy and safety of Cryotherapy combine with Icotinib for Advanced NSCLC Patients harboring EGFR mutation.

DETAILED DESCRIPTION:
In this single arm clinical study, enrolled patients, with advanced stage NSCLC and confirmed epidermal growth factor receptor (EGFR) mutation, would receive cryotherapy for tumors and begin Icotinib, an EGFR tyrosine kinase inhibitor administration thereafter. Progression free survival, overall survival and safety wil be observed.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of non-small cell lung cancer (NSCLC) in phase 3B/4;
* Life expectancy ≥12weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* The number of target lesions in whole body ≤ 8 (and the number of lung lesions ≤ 5, the biggest one's diameter≤ 7 cm, the number of liver lesions ≤ three the biggest one's diameter ≤ 5 cm.
* Adequate hematological function: hemoglobin ≥90g/L (no blood transfusion in 14 days) Absolute neutrophil count (ANC) ≥1.5 * 109/L, and Platelet count ≥75 x 10^9/L.
* Adequate renal function: Serum creatinine ≤1.5 * upper limit of normal(ULN), or Serum creatinine≥ 50 ml/min. Adequate liver function: Total bilirubin ≤ 2 *ULN and Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)< 2.5 * ULN in the absence of liver metastases, or < 5 * ULN in case of liver metastases.
* Female subjects should not be pregnant. All human subjects should able to comply with the required protocol and follow-up procedures, and able to receive oral medications Written informed consent provided.

Exclusion Criteria:

* Previous usage of EGFR-TKI or antibody to EGFR: gefitinib, erlotinib, herceptin, erbitux.
* Allergic to Icotinib.
* Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
* Pregnancy or breast-feeding women.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction with in 6 months, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 2.5 years
  the time that subjects reach their disease progress

SECONDARY OUTCOMES:
overall survival | 3-3.5 years
  the time subjects die

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Liu, M.D., Study Chair — Fuda Cancer Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Govindan R, Page N, Morgensztern D, Read W, Tierney R, Vlahiotis A, Spitznagel EL, Piccirillo J. Changing epidemiology of small-cell lung cancer in the United States over the last 30 years: analysis of the surveillance, epidemiologic, and end results database. J Clin Oncol. 2006 Oct 1;24(28):4539-44. doi: 10.1200/JCO.2005.04.4859. PMID 17008692
- [Background] Zhikai Z, Lizhi N, Liang Z, Jianying Z, Fei Y, Jibing C, Jialiang L, Kecheng X. Treatment of central type lung cancer by combined cryotherapy: experiences of 47 patients. Cryobiology. 2013 Oct;67(2):225-9. doi: 10.1016/j.cryobiol.2013.07.003. Epub 2013 Jul 31. PMID 23911808
- [Background] Shi Y, Zhang L, Liu X, Zhou C, Zhang L, Zhang S, Wang D, Li Q, Qin S, Hu C, Zhang Y, Chen J, Cheng Y, Feng J, Zhang H, Song Y, Wu YL, Xu N, Zhou J, Luo R, Bai C, Jin Y, Liu W, Wei Z, Tan F, Wang Y, Ding L, Dai H, Jiao S, Wang J, Liang L, Zhang W, Sun Y. Icotinib versus gefitinib in previously treated advanced non-small-cell lung cancer (ICOGEN): a randomised, double-blind phase 3 non-inferiority trial. Lancet Oncol. 2013 Sep;14(10):953-61. doi: 10.1016/S1470-2045(13)70355-3. Epub 2013 Aug 13. PMID 23948351